CLINICAL TRIAL: NCT05736497
Title: Integration of Multimodal Cancer Predisposition Genetic Counseling Practices Within the Pediatric Oncology Setting: Digital Care Plans for Patients With CPS
Brief Title: Care Plans for Cancer Predisposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 21-019151; R21HG011912 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Genetic Predisposition
Keywords: genetic testing; genetic counseling; germline testing; digital care plan; cancer predisposition syndrome
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Intervention Model Description: Comparison of pre and post testing of same cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Digital Care Plans with Accompanying Text Messages (Experimental): Investigators will recruit families and patients diagnosed with a Cancer Predisposition Syndrome within 3 years. Participants will be provided with a digital care plan and optional accompanying text message reminders.
  Interventions: Other: Digital Care Plans

INTERVENTIONS:
Other: Digital Care Plans — Investigators will develop digital care plans for 10 common Cancer Predisposition Syndromes for patients diagnosed within 3 years.

SUMMARY:
Develop and evaluate acceptability, feasibility, and preliminary efficacy of digital care plan and accompanying text message reminders for children and adolescents with a known Cancer Predisposition Syndromes (CPS).

DETAILED DESCRIPTION:
As over 15% of pediatric cancers are associated with a cancer predisposition, it is increasingly becoming standard of care for children with cancer, as well as those with suspected hereditary risk, to be evaluated for germline cancer predisposition. Unfortunately, the increase in pediatric genetic testing has exceeded the pace of research supporting effective cancer surveillance in positive cases. Additionally, guidelines for cancer predisposition management are not easily accessed or understood by families; thus, there is often a disconnect between the understanding and retention of such information relayed to families.

In this study, Investigators will develop and evaluate the acceptability, feasibility, and preliminary efficacy of digital care plans for Cancer Predisposition Syndromes (CPS) with accompanying text message reminders for children and adolescents with a known CPS. Digital care plans and text messages will be created for 10 common CPS. Investigators will use a quasi-experimental design with pre and post testing of the same cohort, before and after delivery of care plan and accompanying messages. To evaluate the impact of the digital care plans, Investigators will compare assessments of the same cohorts at 3 and 6 months time points.

ELIGIBILITY:
Inclusion Criteria:

Parents

1. Parent or Legal Guardian of a patient with a known cancer predisposition syndrome diagnosed within the last 5 years
2. Received care at the Cancer Predisposition clinic at the Children's Hospital of Philadelphia (CHOP), or other medical institutions (does not need to be receiving follow-up care at CHOP)
3. Appropriate to approach per oncology team/cancer predisposition team
4. No cognitive impairment limiting ability to complete measures
5. Ability to read and speak English fluently

Adolescent/Young Adult (AYA) probands

1. Child proband with a known cancer predisposition syndrome diagnosed within the last 5 years
2. Ages 12+
3. Received care at the Cancer Predisposition clinic at the Children's Hospital of Philadelphia (CHOP), or other medical institutions (does not need to be receiving follow-up care at CHOP)
4. Appropriate to approach per oncology team/cancer predisposition team
5. No cognitive impairment limiting ability to complete measures
6. Ability to read and speak English fluently

Exclusion Criteria:

* Not meeting any of inclusion criteria

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge Score of participating family members | 3 months and 6 months after receipt of digital care plan
  Change in knowledge score for participating family members will be measured by participants completion of electronic questionnaires administered via REDCap. The change in the mean and standard deviation will be assessed at 3 months and 6 months. A higher score indicates greater knowledge of care plans content.

SECONDARY OUTCOMES:
Acceptability of use of digital care plans for CPS for participating family members | 3 months after receipt of digital care plan
  Acceptability will be measured by participants completion of electronic questionnaires administered via REDCap. Acceptability ratings will be documented with standard descriptive statistics such as means and frequencies. A higher score indicates indicates higher satisfaction, perceived appropriateness, positive effect, demand, and potential for future use.
Feasibility of use of digital care plans for CPS for patients diagnosed within 5 years | Up to 6 months after receipt of digital care plan
  Feasibility will be assessed with absence of technical difficulties allowing the Clinical Research Coordinator (CRC) to create care plan in under 15 minutes in a busy clinical setting.
Satisfaction with decision to have germline testing | Up to 6 months after receipt of digital care plan
  Satisfaction with decision to have germline testing will be measured by participants completion of electronic questionnaires administered via REDCap. The change in the mean and standard deviation will be assessed at 3 months and 6 months and compared to baseline. A higher score indicates greater satisfaction with decision to have child genetically tested.
Change in cancer-related anxiety | Up to 6 months after receipt of digital care plan
  Cancer-related anxiety will be measured by participants completion of electronic questionnaires administered via REDCap. The change in the mean and standard deviation will be assessed at 3 months and 6 months and compared to baseline. A higher score indicates greater cancer-related stress.
Change in distress after receiving genetic test results | Up to 6 months after receipt of digital care plan
  Distress after receipt of genetic test results will be measured by participants completion of electronic questionnaires administered via REDCap. The change in the mean and standard deviation will be assessed at 3 months and 6 months and compared to baseline. A higher score indicates greater distress about genetic test result disclosure.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne MacFarland, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators are committed to making all data, protocols, tools, and materials available to the scientific community, in compliance with Children's Hospital of Philadelphia policies and NIH "Sharing Data and Resources" statement, NIH Grants Policy Statement, and the NIH Office of Extramural Research, Division of Extramural Inventions & Technology Resources (DEITR) Intellectual Property Policy. This includes sharing of protocols freely with collaborators and sharing of data through peer-reviewed publication and presentation in scientific meetings. All members of the research team will comply with the NIH policy on sharing data by protecting the privacy and rights of human subjects involved in the research at all times. All members of the research team with comply with the Health Insurance Portability and Accountability Act of 1996 (HIPAA) and its accompanying regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Upon request

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT05736497/Prot_SAP_000.pdf
  • Informed Consent Form: Written Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05736497/ICF_001.pdf
  • Informed Consent Form: Verbal Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05736497/ICF_002.pdf